CLINICAL TRIAL: NCT00899795
Title: Stromal Injury and Clonal Adaptation in Myelodysplasia
Brief Title: Evaluating Cell Damage in Patients With Acute Myeloid Leukemia, Myelodysplastic Syndromes, or Fanconi Anemia; in Patients Who Were Exposed to Alkylating Agents; and in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Grover Bagby, Professor Emeritus, OHSU Knight Cancer Institute
Other Study IDs: IRB00001025; P30CA069533 (NIH); OHSU-HEM-02008-LX; CDR0000445436 (Other: NCI PDQ)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; untreated adult acute myeloid leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Flow Cytometry; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Other: flow cytometry
Procedure: biopsy

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer and from healthy volunteers in the laboratory may help doctors learn more about changes that occur in bone marrow stromal (connective tissue) cells. It may also help doctors understand the effects of alkylating agents on bone marrow stromal cells.

PURPOSE: This laboratory study is evaluating stromal cells in patients with acute myeloid leukemia, myelodysplastic syndromes, or Fanconi anemia; in patients who were exposed to alkylating agents; and in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine abnormal stromal function in patients with acute myeloid leukemia (AML), myelodysplastic syndromes (MDS), or Fanconi anemia; in patients who were exposed to alkylating agents; and in healthy volunteers.

Secondary

* Determine whether clonal progenitors from patients with secondary AML or MDS are resistant to selected extracellular apoptotic cues.
* Determine whether stromal function in patients with secondary AML or MDS is more aberrant than stromal function in patients with primary AML or MDS.
* Determine whether cytotoxic agents known to induce secondary MDS or AML influence the supportive function of the bone marrow stroma.
* Determine whether cytoprotective agents reduce both cytotoxicity and genotoxicity in hematopoietic progenitor cells and stromal cells.

OUTLINE: Patients and healthy volunteers undergo bone marrow sample collection. Progenitor cells are grown in culture. Cell survival is quantified by flow cytometric and cytogenetic analysis, sister chromatid exchange, and FISH for chromosome 11 changes (for etoposide-exposed samples only).

PROJECTED ACCRUAL: A total of 24 patients and healthy volunteers will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of acute myeloid leukemia or myelodysplastic syndromes and requires bone marrow aspiration/biopsy for clinical purposes

    * Primary or secondary disease
  * Diagnosis of Fanconi anemia by positive mitomycin C test (age 5 to 55 years)
  * Received prior chemotherapy containing any of the following alkylating agents: mechlorethamine, chlorambucil, cyclophosphamide, melphalan, busulfan, or topoisomerase inhibitors
  * Healthy volunteer (age 18 and over), meeting the following criteria:

    * CBC normal
    * WBC > 1,000/mm³
    * Hemoglobin > 10 g/dL
    * Platelet count > 70,000/mm³
* No bone marrow metastases
* No evidence of non-hematopoietic malignancy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* No clinical signs and symptoms of acute or subacute infection (viral, bacterial, or fungal infection)
* No allergy to lidocaine or xylocaine

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 6 months since prior cytotoxic or immunosuppressive agents
* No prior extensive pelvic radiotherapy (> 20 Gy)

Ages: 5 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient, outpatient, and normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2002-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Abnormal stromal function

SECONDARY OUTCOMES:
Clonal progenitors resistant to selected extracellular apoptotic cells
Comparison of stromal function between secondary vs primary acute myeloid leukemia or myelodysplastic syndromes
Influence of cytotoxic agents on supportive function of the bone marrow stroma
Reduction of cytotoxicity and genotoxicity in hematopoietic progenitor cells and stromal cells with use of cytoprotective agents

CONTACTS AND LOCATIONS:
Overall Officials: Grover C. Bagby, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States